CLINICAL TRIAL: NCT03973866
Title: Alfapump® System in the Treatment of Refractory or Recurrent Ascites: a Multicenter Single Arm Within Subject Crossover Design Pivotal Study (the POSEIDON Study)
Brief Title: Alfapump® System in the Treatment of Refractory or Recurrent Ascites (POSEIDON Study)
Acronym: POSEIDON
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sequana Medical N.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-AAR-010
Record Dates: First submitted 2019-05-31; First posted 2019-06-04 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Ascites
MeSH Terms: conditions — Ascites

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Alfapump (Experimental): Implantation of Alfapump
  Interventions: Device: Alfapump

INTERVENTIONS:
Device: Alfapump — Implantation of alfapump

SUMMARY:
The POSEIDON study is a multi-center, prospective, single arm, crossover pivotal study enrolling up to 70 pivotal cohort patients and up to 45 additional Roll-in patients with refractory or recurrent ascites at up to 20 sites. Pivotal cohort patients will undergo a 3-month pre-implant observation phase after enrollment, followed by implantation of the alfapump and 24 months of post-implant follow up. An analysis will be conducted to support an application for device approval when a minimum of 40 treated pivotal cohort patients are through 6 months.

DETAILED DESCRIPTION:
The POSEIDON Study is a multicenter, single arm within subject crossover design pivotal trial conducted in patients diagnosed with refractory or recurrent ascites due to liver cirrhosis who meet inclusion/exclusion criteria. The study will enroll up to 70 pivotal cohort patients with refractory or recurrent ascites at up to 20 sites. In addition, up to 45 additional Roll-in patients will be allowed. An analysis will be conducted to support an application for device approval when a minimum of 40 treated pivotal cohort patients are through 6 months. Patients will be followed for longer-term safety and effectiveness for a total of 2-years post-implant. Patients with a functioning pump at 24 months may consent to continued participation in a long-term follow-up evaluation and with assessments every 3 months from 24 months through the time the pump ceases to function, pump explant or patient death. This long-term follow-up period will continue until the product is approved or the sponsor determines they will no longer pursue product approval.

Pivotal Cohort Patients

Pivotal cohort patients will be evaluated in a 3-month pre-implant observation period during which they will receive standard of care therapy consisting of paracentesis as required for removal of ascitic fluid. Following the initial 3-month observation period during which the number and volume of paracentesis and Quality of life (assessed by general HRQL scores (SF-36)) as well as disease-specific validated questionnaires (Ascites-Q) will be documented, patients will be reevaluated for eligibility for pump implant.

Roll-in Patients

In the study centers without previous experience in pump placement, training in the pump implant procedure will be conducted and up to 3 initial pump implantations conducted as roll-in cases. Roll-in patients will be sequentially enrolled at the site until sufficient experience has been obtained and the site is approved by the sponsor to enroll in the pivotal phase. Roll-in patients will not undergo the 3-month pre-implant observation period and will not be included in the Primary Analysis set but will be summarized separately for purposes of safety evaluation with effectiveness data provided as supplemental. In the event a primary implanter at the site is a replaced or added, up to 3 additional Roll-in implants will be allowed.

All patients (Pivotal and Roll-in) will undergo a final eligibility assessment prior to pump implant. If deemed eligible, patients will be implanted with the alfapump. In the 3 months post-implant, patients will be monitored with pump adjustments as needed to increase or decrease volume of fluid to be removed each day. After this period of stabilization, a 3-month primary endpoint observation period (month 4 through month 6) will begin. In each period, the protocol specifies when symptom driven (therapeutic) paracentesis can be performed per protocol as well as conditions under which the use of diuretics may be considered (all patients must discontinue diuretics post implant procedure).

The study is designed to demonstrate in pivotal cohort patients 1) a 50% reduction (superiority margin) in the per-patient ratio of post-implant 3-month observation period (M4 to M6 post implantation) to pre-implant 3-month observation period with respect to average monthly requirement for therapeutic paracentesis and 2) at least 50% of patients will achieve a 50% reduction in the requirement for therapeutic paracentesis in the same period.

ELIGIBILITY:
Inclusion Criteria:

At the time of Initial Screening:

1. Patients > 18 years of age
2. Cirrhosis of the liver defined by histological and/or clinical, endoscopic, laboratory and radiological criteria.
3. Refractory or recurrent ascites primarily managed with periodic therapeutic paracentesis . Patients must have a minimum of 2 therapeutic paracenteses in the 30 Days prior to enrollment
4. Not a candidate for (e.g. refused, contraindicated) Transjugular intrahepatic portosystemic shunt (TIPS) or previously implanted TIPS is permanently obstructed or non-functioning.
5. Screened for esophageal varices and on optimal management
6. Absence of contraindications to prophylactic antibiotic use from time of pump implant
7. Life expectancy of at least 6 months following pump implant (approximately 10 months from enrollment)
8. Capable of giving written informed consent, willing to comply with study procedures including the 3-month pre-implant observation period and ability to operate and charge the device.
9. Women of childbearing age should use adequate contraceptives.

   Reassessed at time of implant procedure (Pivotal Cohort Only):
10. Has required a minimum of 5 therapeutic paracenteses in the 3-month observation period prior to pump implant

Exclusion Criteria:

At the time of Initial Screening:

1. Renal failure defined as serum creatinine higher than 1.5 mg/dL
2. More than one episode of spontaneous bacterial peritonitis over the previous 6 months
3. More than one episode of bacterascites over the previous 6 months
4. Recurrent urinary infections as per standard criteria, defined as 2 or more episodes over the last 6 months
5. Evidence of loculated ascites, as per imaging
6. Hepatocellular carcinoma, exceeding Milan criteria or for which RF ablation is anticipated
7. Pregnant females or females anticipating pregnancy during study period
8. Patients currently enrolled in another interventional clinical study that has not reached the primary endpoint assessment point, or (for pivotal cohort) patients who have previously had an alfapump implanted
9. Immuno-modulatory treatment (including azathioprine, methotrexate, anti-TNF therapies) used within last 4 months (corticosteroids at stable dose over the last 4 months but < 15 mg/day, or in tapering doses are allowed)
10. Known or suspected hepatic or extra hepatic malignancy (other than skin cancer and in-situ cancers), unless adequately treated or in complete remission for ≥ 3 years
11. History of bladder cancer
12. BMI>40 presenting a risk for technical difficulties for surgery or catheter implantation
13. Contraindications to general anesthesia
14. Comorbid condition or other reason (example hypertension) that may preclude stopping diuretics after enrollment
15. MELD-Na Score > 20
16. Budd Chiari syndrome (Pivotal cohort only)
17. Clostridium difficile infection within the past year

    Assessed or re-assessed at time of pump implant:
18. Acute gastrointestinal hemorrhage requiring transfusions over the previous 42 days
19. Condition that prevents continued cessation of diuretic use
20. Patient condition does not allow the implant procedure to be performed within the limits of acceptable risk (e.g. cardiovascular comorbidities, variceal bleeding within the previous 6 weeks, skin infections or skin ulcers of the anterior abdominal wall within 2 weeks of device placement)
21. Hepatocellular carcinoma exceeding Milan criteria or for which RF ablation is anticipated
22. ICU admission since enrollment in the 30 days preceding pump implant procedure
23. INR >/= 2.0
24. Platelet count of < 50,000 /μL at the time of implantation, unless the platelet count is ≥30,000 / μL and bleeding risk can be satisfactorily addressed with means such as platelet infusion during the implant procedure and/or thrombopoietin receptor agonists
25. Bacterial peritonitis within 4 weeks of implant procedure (this includes peritonitis diagnosed at the time of intervention)
26. Bacterascites within 4 weeks of implant procedure (this includes bacterascites diagnosed at the time of intervention). Note: at the time of final eligibility (just prior to implantation) the subject will not be allowed to move forward with the procedure if he/she has experienced an episode bacterascites within four weeks of the implant procedure date.
27. Serum sodium <125 mmol/L
28. Urinary infection within the last 2 weeks
29. Obstructive uropathy, residual urinary volume exceeding 100 ml, or any bladder anomaly which might contraindicate implantation of the device
30. Evidence of renal failure, defined as serum creatinine higher than or equal to 1.5 mg/dL, in the preceding 30 days
31. Evidence of loculated ascites, as per imaging
32. Pregnant females or females anticipating pregnancy during study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Per-patient ratio of post-implant to pre-implant with respect to average monthly number of therapeutic paracentesis | Comparing data from the post-implant 3-month observation period to data from the pre-implant 3-month observation period:
  Defined as removal of ascites ≥1.5L through needle puncture of abdominal wall
Proportion of patients with at least 50% reduction in number of therapeutic paracenteses from the pre-observation period to post-observation period | Comparing data from the post-implant 3-month observation period to data from the pre-implant 3-month observation period
  Defined as removal of ascites ≥1.5L through needle puncture of abdominal wall
Combined rate of open surgical reintervention due to pump system related adverse event or to restore pump functionality, pump explant due to pump system related adverse event, or pump system related death | from time of pump implant through 6 months post-implant
  Safety of the alfapump implant procedure and alfapump therapy as determined by rates of explant, reintervention, and other serious device or procedure related adverse events

SECONDARY OUTCOMES:
Requirement for large volume paracentesis (LVP): change in the average number of LVP events per month (that consist of removing ≥ 5L of ascitic fluid) | in the post-implant 3-month primary endpoint observation period compared to the pre-implant observation period
  Effectiveness of the alfapump to control ascites as determined by the change in the need for repeated paracentesis compared to baseline
Change of cumulative volume of ascitic fluid removed by means of therapeutic paracentesis | in the post-implant 3-month primary endpoint observation period as compared to the pre-implant 3-month observation period
  Effectiveness of the alfapump to control ascites as determined by the change in the need for repeated paracentesis compared to baseline
Change in SF-36 Physical Component Score | post-implant 3-month primary endpoint observation period as compared to the pre-implant 3-month observation period
  The Medical Outcomes Study Short Form Survey Instrument (SF-36) taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal/emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes one item that indicates a perceived change in health. Scoring the SF-36 is a two-step process. First, precoded numeric values are recoded per a scoring key. A high score defines a more favorable health state. Each item is scored on a 0-100 range. The lowest and highest possible scores are 0 and 100, respectively. Scores represent the percentage of total possible score achieved. In step 2, items in the same scale are averaged together to create the 8 scale scores. Items that are left blank (missing data) are not taken into account when calculating the scale scores. Scale scores represent the average for all items in the scale that the respondent answered.
Change in Ascites-Q Score | in the post-implant 3-month primary endpoint observation period as compared to the pre-implant 3-month observation period
  The Ascites-Q was developed by modifying the Polycystic Liver Disease Questionnaire. It includes 11 out of 16 original questions, covering symptoms of abdominal fullness, anorexia, early satiety, nausea, abdominal pain, back pain, dyspnea, reduced mobility, fatigue, insomnia, discomfort because of abdomen size, and problems with sexual intimacy. One other ascites-specific symptom (insomnia) was added. Each individual symptom is assessed with a frequency (6-point Likert scale "never" to "always") and discomfort (5-point Likert scale "not at all" to "a lot") question. Severity scores of individual symptoms are the sum of the frequency and discomfort score (range 2-11). A higher score represents a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Florence Wong, MD, Principal Investigator — Toronto General Hospital
Locations (15):
- United States (13):
  - Mayo Clinic (Arizona), Phoenix, Arizona
  - Cedars-Sinai Comprehensive Transplant Center, Los Angeles, California
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Duke University, Durham, North Carolina
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Avera Medical Group, Sioux Falls, South Dakota
  - Methodist Dallas, Dallas, Texas
  - Baylor University Medical Center (Dallas), Dallas, Texas
  - McGuire VA Medical Center, Richmond, Virginia
  - Medical College of Wisconsin (Froedtert), Milwaukee, Wisconsin
- Canada (2):
  - Ottawa Hospital, Ottawa, Ontario
  - Toronto General Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wong F, Vagas HE, Reddy KR, Pagadala MR, Pocha C, Sundaram V, Bajaj JS, Shlomovitz E, Bendel E, Capel J, Kamath PS; POSEIDON Study Group. The Effects of Alfapump on Ascites Control and Quality of Life in Patients With Cirrhosis and Recurrent or Refractory Ascites. Am J Gastroenterol. 2025 Oct 1;120(10):2291-2301. doi: 10.14309/ajg.0000000000003300. Epub 2025 Jan 6. PMID 39760647